CLINICAL TRIAL: NCT04703933
Title: Evaluation of the Level of Knowledge and Attitude of the Operating Room Nurses About Radiation Exposure- A Descriptive Study
Brief Title: Knowledge and Attitude of the Operating Room Nurses About Radiation Exposure
Status: Completed | Type: Observational
Sponsor: Acelya Turkmen (Other)
Responsible Party: Sponsor-Investigator, Acelya Turkmen, Research Assistant PhD, Cukurova University
Organization: Cukurova University (Other)
Other Study IDs: 2016-255651
Record Dates: First submitted 2021-01-05; First posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Radiation Exposure; Knowledge, Attitudes, Practice
Keywords: Radiation Protection; Operating Room Nursing; Knowledge; Attitude
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: EVALUATION OF THE LEVEL OF KNOWLEDGE AND ATTITUDE OF THE OPERATING ROOM NURSES — This descriptive study was conducted with 100 nurses working in the operating room of two university hospitals in Istanbul

SUMMARY:
This study aims to evaluate the level of knowledge and attitude of the operating room nurses about radiation exposure.This descriptive study was conducted with 100 nurses working in the operating room of two university hospitals in Istanbul. Descriptive statistical analyses were performed using IBM SPSS 23 (Statistical Package for Social Sciences for Windows, Version 23.00, Armork NY).

DETAILED DESCRIPTION:
Operating rooms are dynamic places where advanced technology is used, and teamwork is best exhibited. Operating room personnel face many biological, physical, and infectious risk factors. One of these risk factors is ionizing radiation. Radiation in the operating room may be spread from non-ionizing devices such as portable X-ray devices and lasers, as well as by radiological methods such as X-ray and fluoroscopy, which have been widely used in recent years as it shortens the duration of surgery.

Radiation is used in many applications in operating rooms and long-term exposure to radiation may occur. Operation room personnel are affected by radiation in three different ways: direct, reflection, and leakage. Influence in the form of leakage is associated with the fluoroscope use and the reflection may occur by transfer from the patient's body or from the objects in the operating room.

Radiation can cause serious adverse effects on hematopoietic, immune, reproductive, circulatory, respiratory, musculoskeletal, endocrine, nervous, digestive, and urinary systems. The negative effects of radiation exposure are generally defined in two ways. The first is acutely occurring determinant effects, and the second is later occurring probabilistic effects. Determinant effects occur as a result of exposure of cells to radiation, in addition to being directly related to cell death. These effects may result in infertility, cataract, leukemia, skin burns, and death. Probabilistic effects are associated with the absorption of radiation accumulated in tissues and may occur even at the lowest dose. Genetic disorders and cancer formation are some of the consequences of probabilistic effects.

The use of protective equipment has a very important role in reducing radiation exposure. The use of masks ensures protection from respiratory hazards, the use of protective clothing ensures that the radioactive substance does not damage the skin and hair, and the use of personal dosimeters ensures the management of the duration of stay in an area with high radiation levels and the monitoring of accumulated doses. Accordingly, the radiation exposure of the operating room nurses is very high. Therefore, nurses should have sufficient information about radiation and protection from radiation. This study was carried out to evaluate the knowledge level and attitude of operating room nurses about radiation exposure.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65 years
* Working in the operating room
* Using the scopy
* Working in the operating room for at least 1 month

Exclusion Criteria:

* Working in a unit other than the operating room
* Working in the operating room for less than a month
* Not using scopy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The research was carried out in two university hospitals in Istanbul. The sample of the study consisted of 100 volunteer operating room nurses.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Knowledge of the Operating Room Nurses About Radiation Exposure | an average of 6 month
  Evaluation of the level of knowledge was done "Data Collection Form" developed by the researcher. The questionnaire consisted of a total of 18 questions.
Attitude of the Operating Room Nurses About Radiation Exposure | an average of 6 month
  Evaluation of the level of attitude was done "Data Collection Form" developed by the researcher. The questionnaire consisted of a total of 18 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Ayfer OZBAS, PhD, Prof., Study Director — Istanbul University - Cerrahpasa; Acelya TURKMEN, PhD, Study Chair — Cukurova University; Gönül YILMAZ DUNDAR, PhD, Study Chair — Bandırma 17 Eylul University

IPD SHARING:
Plan to Share IPD: No